CLINICAL TRIAL: NCT00216853
Title: A Study of Vaginal MicroFlora and Immune Profiles of Patients With Recurrent Urinary Tract Infection
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Dr S. Pautler, Lawson Health Research Institute
Other Study IDs: R-03-202; 9875E
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2009-04-16 (Estimated); Status verified 2009-04

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with Recurrent UTI
- Healthy controls

SUMMARY:
The purpose of this study is to determine the extent to which vaginal microflora and immune profiles of patients with urinary tract infection (UTI) differ from healthy controls.

DETAILED DESCRIPTION:
Recurrent urinary tract infections, which occur mostly in the female population, can be potentially harmful if not treated and significantly reduce quality of life. By characterizing the vaginal microflora and immune profiles of women that suffer recurrent UTIs in contrast to a healthy age matched normal group of women (with no history of recurrent UTIs), we can better understand the differences. This in turn can lead to development of better quality probiotics that will be based on their scientific basis, clinical efficacy, and quality in terms of shelf life and delivery to target sites. The reduction in only one third of UTI cases seen each year would have a significant impact on reducing health care costs.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for UTI Group:

1. At least 2 recurrent UTIs within the last year
2. Written informed consent

Inclusion Criteria for Normal Group:

1. No UTI within the past 5 years
2. Written informed consent

Exclusion Criteria:

Exclusion Criteria for Both Groups:

1. Active UTI
2. Urinary tract anomalies
3. Evidence of a neurogenic bladder
4. Known immunodeficiencies
5. Use of antibiotics, within the last month
6. Concomitant use of oral steroids
7. Known renal calculi
8. Previous or ongoing chemotherapy
9. Pregnancy

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2003-09; Primary Completion 2006-06 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Pautler, MD, FRCSC, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- St. Joseph's Health Centre, London, Ontario, Canada